CLINICAL TRIAL: NCT03652571
Title: Tailored Treatment of Functional Dyspepsia With Nortriptyline: a Multi-center Double-blind Placebo-controlled Trial
Brief Title: Nortriptyline for the Treatment of Functional Dyspepsia
Acronym: TENDER
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The inclusion of participants went more difficult than initially thought. Preliminary analysis showed that the difference between the groups was great enough to draw conclusions from it, so the trial is terminated prematurely.
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 848016005; NL62932.068.17 / METC173051 (Other: METC azM/UM); 2017-003307-21 (EudraCT Number)
Record Dates: First submitted 2018-08-17; First posted 2018-08-29 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2018-08

CONDITIONS: Functional Dyspepsia
MeSH Terms: interventions — Nortriptyline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nortriptyline (Experimental): Nortriptyline in an escalating dose regimen:
  Week 1-2: 10mg daily Week 3-4: 25mg daily Week 5-12: 50mg daily
  Interventions: Drug: Nortriptyline
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nortriptyline — Nortriptyline escalating dose regimen:
  Week 1-2: 10mg Week 3-4: 25mg Week 5-12: 50mg
  Arms: Nortriptyline
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Functional dyspepsia (FD) is a common functional gastrointestinal disorder characterized by upper abdominal discomfort/pain and/or symptoms of meal-related fullness/satiety. There is currently no definitive therapy that is beneficial for all FD patients. Accumulating evidence suggests efficacy of tricyclic antidepressants (TCAs) in FD. However, no firm conclusion can be drawn currently due to the relatively small amount of studies and large heterogeneity between studies. In addition, TCAs are often associated with side effects, which occur early after initiation of therapy preceding the therapeutic effect and often result in discontinuation of the therapy. These side effects are related to drug metabolism, which depend on polymorphisms of the cytochrome P (CYP) enzyme system. It is therefore hypothesized that pre-treatment assessment of CYP genotype and subsequent exclusion of abnormal metabolizers limits the occurrence of side-effects and as such improves compliance and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years;
* A diagnosis of FD according to the Rome IV criteria;
* Predicted CYP2D6 extensive metabolizer phenotype on the basis of CYP genotyping
* Insufficient effect of first line treatment with proton pump inhibitors (twice daily) or prokinetics;
* In the presence of alarm symptoms, patients are required to have undergone an upper gastrointestinal endoscopy (without evidence of organic disease), and have tested negative for Helicobacter pylori 2 years prior to inclusion;
* Women in their fertile age (<55 years old) must use contraception or be postmenopausal for at least two years.

Exclusion Criteria:

* Predicted CYP2D6 poor, intermediate or ultrarapid metabolizer phenotype on the basis of CYP genotyping
* Evidence of current anxiety and/or depression disorder as defined by a score ≥ 10 on the GAD-7 and/or PHQ-9 questionnaire;
* Current use or any previous use of psychotropic medication in the last 3 months prior to inclusion;
* Inability to discontinue prokinetics, NSAIDs or opioids;
* Using drugs of abuse;
* Using more than 2 or 3 units of alcohol per day (females and males respectively)
* Previous major abdominal surgery or radiotherapy interfering with gastrointestinal function:

  1. Uncomplicated appendectomy, cholecystectomy and hysterectomy allowed unless within the past 6 months;
  2. Other surgery upon judgment of the principle investigator;
* History of gastric ulcer;
* History of liver disease, cholangitis, achlorhydria, gallstones or other diseases of the gallbladder/biliary system;
* History of epilepsy
* History of glaucoma
* Pregnancy or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Symptom response | 12 weeks
  Response to therapy, as defined by a 30% reduction from baseline (i.e. the run-in period) in the weekly average of daily symptom scores, during at least 50% of weeks 3-12 of treatment. Symptoms will be assessed daily using a digital diary (mobile phone application). Recorded symptoms include the five core symptoms of FD: epigastric pain, epigastric burning, postprandial fullness, early satiety and upper abdominal bloating.

SECONDARY OUTCOMES:
Adequate relief | 12 weeks
  Self-reported adequate relief. Adequate relief is defined as a 'yes' response in at least 50% of weeks 3-12 of the treatment. Reported via digital diary (mobile phone application)
General quality of life | 12 weeks, 3 & 6 months
  Assessed with the use of the Euro-Qol-5D (EQ-5D; change from baseline).
Dyspepsia-specific quality of life | 12 weeks, 3 & 6 months
  Dyspepsia-specific quality of life, assessed with the use of the Nepean Dyspepsia Index (NDI; change from baseline).
Cost-utility | 12 weeks, 3 & 6 months
  Cost-utility, as determined by calculations incorporating total treatment costs and changes in EQ-5D-5L (QALYs gained), and results from the Medical Consumption Questionnaire (MCQ) and Productivity Cost Questionnaire (PCQ) [savings from reduced medical resource use and increased work productivity respectively].
Use of rescue medication. | 12 weeks
  As reported via digital diary (mobile phone application)
Number and severity of side effects. | 12 weeks
  As reported via digital diary (mobile phone application)
Responder rates following discontinuation | 6 months
  Responder rates following discontinuation of treatment at 6 months follow-up, as defined by a "Yes" to the query regarding adequate relief from baseline symptoms.
Negative mood - anxiety | 12 weeks, 3 & 6 months
  Assessed with the use of the Generalized Anxiety Disorder-7 (GAD-7; change from baseline)
Negative mood - depression | 12 weeks, 3 & 6 months
  Assessed with the use of the Patient Health Questionnaire-9 (PHQ-9; change from baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Ad A.A.M Masclee, Prof, Principal Investigator — Maastricht University Medical Center
Locations (14):
- Netherlands (14):
  - Jeroen Bosch ziekenhuis, 's-Hertogenbosch
  - AMC, Amsterdam
  - VUmc, Amsterdam
  - Rijnstate, Arnhem
  - Gelderse Vallei, Ede
  - Medisch Spectrum Twente, Enschede
  - Martini Ziekenhuis, Groningen
  - Tergooi Hilversum, Hilversum
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Alrijne ziekenhuis, Leiden
  - Maastrich University Medical Center, Maastricht
  - Bernhoven, Uden
  - Diakonessenhuis, Utrecht
  - MMC, Veldhoven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bosch DH, Beckers AB, Snijkers JTW, Bosman MH, Winkens B, Muris JWM, de Wit N, Brouwers JR, van Hee K, Clemens CHM, Haarhuis BJT, Witteman BJM, Masclee AAM, Keszthelyi D. Tailored treatment of functional dyspepsia with nortriptyline: a multi-center, double-blind, placebo-controlled trial. Clin Gastroenterol Hepatol. 2026 Jan 28:S1542-3565(26)00041-8. doi: 10.1016/j.cgh.2026.01.013. Online ahead of print. PMID 41616902